CLINICAL TRIAL: NCT05022888
Title: Investigation of the Diagnostic Effect of Muscle Tissue Oxygenation Values in Patients With Myofascial Pain Syndrome
Brief Title: Near-Infrared Spectroscopy in Myofascial Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. Burcu Metin Ökmen, Principal Investigator ,Assoc. PhD. M.D., Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BYIERH3
Record Dates: First submitted 2021-08-21; First posted 2021-08-26 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Myofascial Pain Syndrome; Regional Tissue Oxygen Saturation
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Intervention Model Description: prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- myofascial pain syndrome (Active Comparator): Patients diagnosed with myofascial pain syndrome Tissue oxygen saturation measured from 4 different regions defined on the trapezius muscle
  Interventions: Device: regional tissue saturation
- Healthy volunteers (Active Comparator): Healthy volunteers Tissue oxygen saturation measured from 4 different regions defined on the trapezius muscle
  Interventions: Device: regional tissue saturation

INTERVENTIONS:
Device: regional tissue saturation — tissue oxygen saturation measured from 4 different regions defined on the trapezius muscle. The NIRS probe will be used in these areas.

SUMMARY:
Myofascial pain syndrome is a regional pain syndrome accompanied by sensorial, motor and autonomic symptoms . myofascial trigger points are most frequently detected in the upper trapezius, levator scapula, and axial postural muscles such as rhomboid major. Myofascial pain syndrome is characterized by active myofascial trigger points in the form of focal hyperirritable nodules palpated in the tight band of the muscle .

Alteration of tissue vascularization could limit or prevent th may cause adhesions, contractures and pain. As a result of decreased blood flow, tissue oxygenation may decrease.

DETAILED DESCRIPTION:
In this study, it will be tried to determine the role of muscle tissue oxygenation in the activity and diagnosis of the disease in myofascial pain syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* myofascial pain syndrome

Exclusion Criteria:

* Cervical radiculopathy
* Fibromyalgia
* Shoulder joint disease,
* Peripheral and central nervous system disease
* Polyneuropathy,
* Inflammatory rheumatic disease,
* Malignancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-23 (Estimated); Primary Completion 2021-11-23 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
regional tissue saturation | 15 minute
  tissue oxygen saturation measured from 4 different regions defined on the trapezius muscle. The NIRS probe will be used in these areas.

SECONDARY OUTCOMES:
peripheral oxygen saturation | 15 minute
  A pulse oximeter will be used to measure peripheral oxygen saturation
Visual Analogue Scale (VAS) | 6 month
  for pain. 0: no pain at all, 10: worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Burcu M.D Metin ÖKMEN, Assoc. PhD., Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital; Korgün MD Ökmen, Assoc. PhD., Study Chair — Bursa Yuksek Ihtisas Training and Research Hospital